CLINICAL TRIAL: NCT07265440
Title: The Efficacy of Effleurage Massage on Striae Gravidarum During Pregnancy
Brief Title: Effect of New Specialized Technique Using Effleurage Massage on Striae Gravidarum
Acronym: EM/SG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Eman Khaled Mohamed Fathelbab, Senior physical therapist in physical therapy for woman health Department, Sidi-Salem Hospital, Kafrelsheikh, Egypt, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KFSIRB200-764
Record Dates: First submitted 2025-11-22; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Striae Gravidarum
MeSH Terms: conditions — Striae Distensae

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Efficacy of EM on SG (Active Comparator): Each patient in this group will perform effleurage massage in transverse direction from medial to lateral only not back and forth, twice a day starting from the 17th week until the 28th week of pregnancy and three times a day starting from the 28th week of pregnancy for 10 minutes for each time until date of birth but from lateral to medial. It will be performed on the whole abdominal area extending from the diaphragm to the pupic area, also on both sides of the abdomen extending from the 12th rib to the iliac crest.
  Interventions: Other: New specialized technique using effleurage massage
- Efficacy of olive oil only on SG (Active Comparator): They will apply olive oil only twice a day starting from the 17th week until the 28th week of pregnancy and three times a day starting from the 28th week of pregnancy until date of birth .
  Interventions: Other: New specialized technique using effleurage massage

INTERVENTIONS:
Other: New specialized technique using effleurage massage — effleurage massage was performed in transverse direction from medial to lateral only not back and forth, twice a day starting from the 17th week until the 28th week of pregnancy and three times a day starting from the 28th week of pregnancy for 10 minutes for each time until date of birth but from lateral to medial. It will be performed on the whole abdominal area extending from the diaphragm to the pupic area, also on both sides of the abdomen extending from the 12th rib to the iliac crest.

SUMMARY:
The goal of this clinical trial is to learn if our new specialized technique using effleurage massage works to prevent striae gravidarum in primigravida. The main questions it aims to answer are:

Can our new specialized technique using effleurage massage prevent or even decrease the severity of striae gravidarum in primigravida ? What side effects may participants face when using our technique?

Participants will:

perform effleurage massage in transverse direction from medial to lateral only not back and forth, twice a day starting from the 17th week until the 28th week of pregnancy and three times a day starting from the 28th week of pregnancy for 10 minutes for each time until date of birth but from lateral to medial. It will be performed on the whole abdominal area extending from the diaphragm to the pupic area, also on both sides of the abdomen extending from the 12th rib to the iliac crest.

DETAILED DESCRIPTION:
This study will be conducted to investigate if our new specialized technique using effleurage massage can prevent or even decrease the severity of striae gravidarum in primigravida .

Participants will:

perform effleurage massage in transverse direction from medial to lateral only not back and forth, twice a day starting from the 17th week until the 28th week of pregnancy and three times a day starting from the 28th week of pregnancy for 10 minutes for each time until date of birth but from lateral to medial. It will be performed on the whole abdominal area extending from the diaphragm to the pupic area, also on both sides of the abdomen extending from the 12th rib to the iliac crest.

ELIGIBILITY:
Inclusion Criteria:

* • All females will be primigravida.

  * All females will be at the 17th week to the 20th week of gestation.
  * Age of participants will range from 20-30 years.
  * Their BMI will not exceed 28 kg/m.

Exclusion Criteria:

* • Any dermal pathology.

  * Psychiatric disorders.
  * Skin tumor.
  * Pregnant with more than one child.
  * History or symptoms of premature birth.
  * Placental abruption.
  * History of abdominal surgeries.
  * History of abdominal hernia.

Ages: 20 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 42 (Actual)
Dates: Start 2024-10-09 (Actual); Primary Completion 2025-01-12 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Reduction in Striae Gravidarum severity | At 21 weeks of gestation, 29 weeks of gestation ,and 39 weeks of gestation
  Severity of striae gravidarum will be assessed using INA score at three time points during pregnancy to evaluate progression and response to the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient Clinics, Faculty of Physical Therapy, Kafrelsheikh University, Egypt, Kafr ash Shaykh, Kafr el-Sheikh Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. This study involves sensitive participant information and there is no plan for data sharing.